CLINICAL TRIAL: NCT02501317
Title: Scientific Validation of the "Active Perineal Rehabilitation" Protocol to Urinary Incontinence Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Laira Lopes Ramos, Master, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 435522
Record Dates: First submitted 2015-07-10; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; physical therapy; rehabilitation; pelvic floor; perineum; conservative treatment
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Perineal Rehabilitation protocol (Experimental): study group that will be treated with "Active Perineal Rehabilitation" protocol
  Interventions: Behavioral: Active Perineal Rehabilitation protocol
- Kari Bo protocol (Active Comparator): control group will be treated with the protocol already widely used
  Interventions: Behavioral: Kari Bo protocol

INTERVENTIONS:
Behavioral: Active Perineal Rehabilitation protocol — Active Perineal Rehabilitation Protocol available in http://www.perineo.info/wordpress/book-active-perineal-rehabilitation/
  Arms: Active Perineal Rehabilitation protocol
Behavioral: Kari Bo protocol — Group exercises to pelvic floor rehabilitation
  Arms: Kari Bo protocol

SUMMARY:
Introduction: Urinary incontinence is a condition that affects most women in her adult life; it is considered a public health problem and has a high negative impact on the quality of life. Physical therapy is considered as the first treatment option for this disease, these treatments are done with pelvic floor muscles exercises (kinesiotherapy) with or without the use of other resources such as biofeedback, electrical stimulation and vaginal cones. Rationale: The protocols used in the various studies on the treatment of urinary incontinence are made with only one type of therapy and have no change in the intensity of the exercises. The "Active Perineal Rehabilitation" protocol uses kinesiotherapy with biofeedback, electrical stimulation, vaginal cones and home exercises; it consists of 14 individual sessions that gradually evolve the intensity of exercises. Objective: To assess the scientific validity of "Active Perineal Rehabilitation" protocol for the treatment of urinary incontinence. Methodology: A multicenter, prospective clinical trial, controlled and randomized, the sample will be divided into a study group that will be treated with the Active Perineal Rehabilitation protocol, and a control group will be treated with the protocol already widely used.

Keys Words: urinary incontinence, physical therapy, rehabilitation, pelvic floor, perineum, conservative treatment

DETAILED DESCRIPTION:
Urinary incontinence is defined as an involuntary loss of urine, the World Health Organization (WHO) considers it is a public health problem having a negative impact on the quality of life of such patients. Its prevalence ranges from 3% to 55%, it is difficult to have a right number because different definitions used and the range age of the population studied. Its more common type is stress urinary incontinence (SUI), the involuntary loss of urine on exertion, coughing or sneezing.

In the old days, those pathologies were seen as a natural consequence of aging, making people adapt to the changes imposed by them. Modern society and the increase of life expectancy made people care more about their quality of life and well-being, making them search for treatments to those pathologies.

The International Federation of Gynecology and Obstetrics, International Continence Society, as well the most of national societies of gynecology and urology, deliberate that physiotherapy is the first option to urinary incontinence treatment. Perineal rehabilitation aims increase pelvic floor muscle strength, to intensify urethral closure.

Perineal rehabilitation is showing to be an efficient treatment to urinary incontinence, studies show that rate cure is between 28 to 84%, this large interval is because different techniques and different assessments in each study.The treatments used in perineal rehabilitation are kinesiotherapy (pelvic floor muscle exercises), with or without biofeedback, electrical stimulation and vaginal cones.

Although there are several studies about physical therapy to urinary incontinence treatment, there are not studies that use more than one of these techniques. Other problem is the fact that the protocols used in these studies start and finish with the same exercises intensity, there is no evolution in the treatment. It can be observed in the literature review made by Hay-Smith, 2012 and Margarida Ferreira e Paula Santos, 2011.

The "Active Perineal Rehabilitation" (APR) protocol uses perineal kinesiotherapy with biofeedback, electrical stimulation, vaginal cones and home exercises, its intensity increase session by session, like is recommended by American College of Sports Medicine. This protocol is unique and innovative to urinary incontinence treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosticated with stress urinary incontinence, with stress test positive; and age between 20 to 75 years old.

Exclusion Criteria:

* Pregnancy
* Metallic intrauterine device
* Unable to understand physical therapist orientations
* Urinary infection
* Virginity
* Prolapse grade 2 or more
* Previous pelvic surgery
* Previous treatment to urinary incontinence in the last 6 months before the study

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Urinary loss frequency | 6 months
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form and stress test

SECONDARY OUTCOMES:
Quality of life | 6 months
  Incontinence quality of life questionnaire
Sexual satisfaction | 6 months
  Female sexual function index

CONTACTS AND LOCATIONS:
Overall Officials: Laira Ramos, master, Principal Investigator — Federal University of São Paulo